CLINICAL TRIAL: NCT03303313
Title: A Phase 2, Open Label, Multicenter Study of ALN-CC5 Administered Subcutaneously in Adult Patients With Atypical Hemolytic Uremic Syndrome
Brief Title: A Study of an Investigational Drug, Cemdisiran (ALN-CC5), in Patients With Atypical Hemolytic Uremic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to lack of enrollment.
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-CC5-004
Record Dates: First submitted 2017-09-25; First posted 2017-10-06 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: RNAi therapeutic; Atypical Hemolytic Uremic Syndrome; Hemolysis; Thrombocytopenia; Renal insufficiency; Thrombotic Microangiopathy; aHUS; TMA
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Hemolysis; Thrombocytopenia; Renal Insufficiency; Thrombotic Microangiopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cemdisiran (Experimental)
  Interventions: Drug: Cemdisiran

INTERVENTIONS:
Drug: Cemdisiran — Subcutaneous (sc) injection of Cemdisiran

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of Cemdisiran in patients with aHUS.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent and to comply with the study requirements
2. Age 18 years or older
3. Clinical diagnosis of primary aHUS
4. Clinical thrombotic microangiopathy (TMA) activity
5. Women of child-bearing potential must have a negative pregnancy test, cannot be breast feeding, and must be willing to use a highly effective method of contraception
6. Previously vaccinated with meningococcal group ACWY conjugate vaccine and meningococcal group B vaccine or willingness to receive these vaccinations
7. ADAMTS13 >10% or other proven aHUS-associated mutation

Exclusion Criteria:

1. Clinically significant abnormal laboratory results
2. Positive Shiga toxin producing Escherichia coli test at Screening
3. Suspected secondary aHUS, in the opinion of the Investigator (unless there is a documented aHUS-associated genetic mutation)
4. Positive direct Coombs test
5. Patients who have received hemodialysis for >3 months
6. Bone marrow transplant recipients
7. Organ transplant recipients, except for kidney transplant recipients with primary aHUS (confirmed by known genetic mutation and kidney biopsy)
8. Known history or evidence of systemic lupus erythematosus or antiphospholipid antibody syndrome
9. History of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc
10. Malignancy (except for non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma) within the last 5 years
11. Patients with a poor prognosis that is expected to limit their life expectancy to less than 3 months, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
The effect of Cemdisiran on platelet count | Week 32

SECONDARY OUTCOMES:
The effect of Cemdisiran on hematological response as measured by platelet count | after 32 weeks of treatment
The effect of Cemdisiran on hematological response as measured by lactate dehydrogenase (LDH) | after 32 weeks of treatment
The effect of Cemdisiran on hematological response as measured by rescue plasma therapy | after 32 weeks of treatment
The effect of Cemdisiran on LDH response as measured by LDH | after 32 weeks of treatment
The effect of Cemdisiran on LDH response as measured by rescue plasma therapy | after 32 weeks of treatment
The effect of Cemdisiran on complete Thrombotic microangiopathy (TMA) response as measured by platelet count | after 32 weeks of treatment
The effect of Cemdisiran on complete Thrombotic microangiopathy (TMA) response as measured by LDH | after 32 weeks of treatment
The effect of Cemdisiran on complete Thrombotic microangiopathy (TMA) response as measured by serum creatinine levels | after 32 weeks of treatment
The effect of Cemdisiran on complete Thrombotic microangiopathy (TMA) response as measured by rescue plasma therapy | after 32 weeks of treatment
The effect of Cemdisiran on serum creatinine levels | up to 84 weeks
The effect of Cemdisiran on estimated glomerular filtration rate (eGFR) | up to 84 weeks
The effect of Cemdisiran on adverse events (AEs) | up to 108 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nader Najafian, MD, Study Director — Alnylam Pharmaceuticals
Locations (12):
- Clinical Trial Site, Sarajevo, Bosnia and Herzegovina
- Clinical Trial Site, Calgary, Canada
- Estonia (2):
  - Clinical Trial Site, Tallinn
  - Clinical Trial Site, Tartu
- Clinical Trial Site, Tbilisi, Georgia
- Clinical Trial Site, Riga, Latvia
- Lithuania (2):
  - Clinical Trial Site, Kaunas
  - Clinical Trial Site, Vilnius
- Clinical Trial Site, Chisinau, Moldova
- Clinical Trial Site, Skopje, North Macedonia
- Clinical Trial Site, Belgrade, Serbia
- Clinical Trial Site, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided